CLINICAL TRIAL: NCT03524807
Title: Effect of Pelvic Floor Muscle Electrophysiologic Therapy on Enhanced Recovery After Gynecologic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, chief physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: electrophysiologic treatment
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Pelvic Floor Muscle Electrophysiologic Therapy; Fast-Track Surgery
Keywords: pelvic floor muscle electrophysiologic therapy; enhanced recovery; muscle soreness; postoperative retention of urine; Intrauterine Adhesions; enhanced recovery after gynecologic surgery
MeSH Terms: conditions — Myalgia; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrophysiologic therapy group (Experimental): apply electrophysiologic therapy after surgery
  Interventions: Device: Electrophysiologic therapy
- non-electrophysiologic therapy group (No Intervention): do not apply electrophysiologic therapy after surgery

INTERVENTIONS:
Device: Electrophysiologic therapy — Pelvic floor electrophysiological therapy is used after common gynecologic surgery to record anal exhaust time and micturition time after surgery and endometrium recovery of intrauterine adhesions.For intrauterine adhesions patients, Drug: Aspirin(low dose of Aspirin after operation)Device: intrauterine balloon (insert intrauterine balloon after operation)
  Other Names: pelvic floor muscle electrophysiologic therapy
  Arms: Electrophysiologic therapy group

SUMMARY:
This study is to evaluate the effect of pelvic floor muscle electrophysiologic therapy on enhanced recovery after gynecologic surgery,to solve muscle soreness and retention of urine after laparoscopy, and endometrial repair after electrosurgical resection of intrauterine adhesions.

DETAILED DESCRIPTION:
Pelvic floor muscle electrophysiologic therapy is widely used in the treatment of pelvic floor dysfunction diseases at home and abroad. Electrical stimulation can also relieve depression and anxiety and play a sedative effect. In recent years, some studies have shown that pelvic floor electrophysiological therapy can improve the intimal blood flow resistance index of thin endometrium. Therefore, whether or not the pelvic floor electrophysiological therapy can relieve the muscle soreness caused by carbon dioxide retention after endoscopic surgery, reduce the postoperative urinary retention, shorten the postoperative anus exhaust time, and repair the endometrium after the intrauterine adhesion. we expect this electrophysiologic therapy can solve some common postoperative complications and difficult problems, such solve muscle soreness and retention of urine after laparoscopy, and endometrial repair after electrosurgical resection of intrauterine adhesions. Hope to help patients recover quickly after surgery.

ELIGIBILITY:
Inclusion Criteria:

.After electrocision of intrauterine adhesions;

.Or after common gynecologic laparoscopic surgery，patients occurred muscle pain or patients occurred urinary retention.

Exclusion Criteria:

* Pregnancy;
* Suspected acute inflammation of the genitourinary system;
* Postoperative persistent vaginal bleeding;
* Patients have vaginal stenosis;
* Patients have implantation of a pacemaker with a cardiac pacemaker;
* Patients have a malignant pelvic organ tumor; .Patients have nervous system disease (dementia or unstable seizures),who cannot actively cooperate with the treatment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
time of anal exhaust and urination after gynecologic surgery | within three days after gynecologic surgery
Endometrial Thickness of All Participants in the Mid Menstrual Measured by Color Doppler Ultrasound | Within the first 3 months after surgery

SECONDARY OUTCOMES:
Menstruation Pattern(Improvement or No Significant Change) of All Participants | Within the first 3 months after surgery
Reduction of American Fertility Society adhesion score at Second-look hysteroscopy of All Participants | Within the first 3 months after surgery
  The severity and extent of intrauterine adhesions were scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version) [7]. A score of 1-4 was considered to represent mild adhesions, a score of 5-8 was considered to represent moderate adhesions and a score of 9-12 represented severe adhesion
Number of Participants With Pregnancy after operation | within three years

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Chen, Chief, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China